CLINICAL TRIAL: NCT02234115
Title: An Open-Labeled, Singled-Arm Study of the Safety, Efficacy, and Pharmacokinetic Behavior of Leuprolide Mesylate for Injectable Suspension (LMIS 50 mg) in Subjects With Advanced Prostate Carcinoma
Brief Title: Safety, Efficacy, and Pharmacokinetic Behavior of Leuprolide Mesylate in Subjects With Advanced Prostate Carcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Foresee Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FP01C-13-001; 2013-001790-25 (EudraCT Number)
Record Dates: First submitted 2014-09-01; First posted 2014-09-09 (Estimated); Results first posted 2018-04-13 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Prostatic Neoplasms
Keywords: Prostate Neoplasm Cancer Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Leuprolide Mesylate 50mg (Experimental): All subjects will be males with advanced prostate carcinoma. They will be injected twice with a depot formulation containing 50 mg of Leuprolide Mesylate. The first dose on day 0 the second dose on day 168 (six months apart). Subjects will be followed until day 336.
  Interventions: Drug: Leuprolide Mesylate

INTERVENTIONS:
Drug: Leuprolide Mesylate — Subcutaneous injection of 50mg Leuprolide Mesylate

SUMMARY:
The study will evaluate if Leuprolide Mesylate is safe and effective in the treatment of subjects with advanced prostate carcinoma, when administered as two injections six months apart.

DETAILED DESCRIPTION:
This is a multi-center, open-label, single-arm study conducted in 2 parts. Part I was established to provide a vanguard of the first 30 subjects who will have more frequent monitoring of their safety. If safety is established, the remainder of the subjects will be entered into the clinical study (i.e., Part II). All subjects will be males with advanced prostate carcinoma judged to be candidates for medical androgen ablation therapy, and all will receive two injections of LMIS 50 mg six-month apart in an unblinded fashion.

ELIGIBILITY:
Inclusion Criteria:

1. Males aged ≥ 18 years old
2. Males with histologically confirmed carcinoma of the prostate
3. Subjects who are judged by the attending physician and/or Principal Investigator to be a candidate for androgen ablation therapy
4. Baseline morning serum testosterone level > 150 ng/dL performed at Screening Visit
5. Eastern Cooperative Oncology Group (ECOG) Performance score ≤ 2
6. Life expectancy of at least 18 months
7. Laboratory values

   * Absolute neutrophil count ≥ 1,500 cells/µL
   * Platelets ≥ 100,000 cells/µL
   * Hemoglobin ≥ 10 gm/dL
   * Total bilirubin ≤ 1.5 × upper limit of normal (ULN)
   * AST (SGOT) ≤ 2.5 × ULN
   * ALT (SGPT) ≤ 2.5 × ULN
   * Serum creatinine ≤ 1.5 mg/dL
   * Lipid profile within acceptable range according to investigator's judgment
   * HgbA1c within acceptable range according to investigator's judgment
   * Clinical chemistries (K, Na, Mg, Ca and P) within acceptable range according to investigator's judgment
   * Serum glucose within acceptable range according to investigator's judgement
   * Urinalysis within normal range according to the investigator's judgment
8. Agree to use male contraceptive methods during study trial
9. Based on the Investigator's judgment, the ability to understand the nature of the study and any hazards of participation, and to communicate satisfactorily with the Investigator and to participate in, and to comply with, the requirements of the entire protocol
10. All aspects of the protocol explained and written informed consent obtained

Exclusion Criteria:

* Receipt of chemotherapy, immunotherapy, cryotherapy, radiotherapy, or anti- androgen therapy concomitantly, or within 8 weeks prior to Screening Visit, for treatment of carcinoma of the prostate. Radiation for pain control will be allowed during the study.
* Receipt of any vaccination (including influenza) within 4 weeks of Baseline
* History of blood donation within 2 months of Baseline
* History of anaphylaxis to any LH-RH analogues
* Receipt of any LHRH suppressive therapy within 6 months of Baseline
* Major surgery, including any prostatic surgery, within 4 weeks of Baseline
* History and concomitant clinical and radiographic evidence of central nervous system/spinal cord metastases. Subjects at risk for spinal cord compression will be excluded.
* Clinical evidence of active urinary tract obstruction and subjects at risk for urinary obstruction
* History of bilateral orchiectomy, adrenalectomy, or hypophysectomy
* History or presence of hypogonadism, or receipt of exogenous testosterone supplementation within 6 months of Baseline
* Clinically significant abnormal ECG and/or history of clinically significant cardiovascular disease as judged by the investigator
* History of drug and/or alcohol abuse within 6 months of Baseline
* Contraindication to leuprolide or an LHRH agonist as indicated on package labeling
* Use of 5-alpha reductase inhibitor within the last 6 months of Baseline
* History or presence of insulin-dependent diabetes mellitus (Type I). Presence of well controlled diabetes mellitus Type II will be allowed
* Use of systemic corticosteroids at a dose >10 mg/d or anti-androgens
* Use of any investigational agent within 4 weeks of Baseline
* Use of any over-the-counter (OTC) medication within 4 weeks of Baseline except for those listed in the permitted Concomitant Treatment section.
* Uncontrolled intercurrent illness that would jeopardize the subject's safety, interfere with the objectives of the protocol, or limit the subject's compliance with study requirements, as determined by the Investigator in consultation with the Sponsor

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2014-08; Primary Completion 2016-08-30 (Actual); Study Completion 2017-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Mao, PhD, Study Director — Foresee Pharmaceuticals Co., Ltd.
Locations (29):
- United States (8):
  - Urology Centers of Alabama, Homewood, Alabama
  - Alliance Research Centers, Laguna Hills, California
  - Genesis Research, LLC, San Diego, California
  - Idaho Urologic Institute - Meridian, Meridian, Idaho
  - AdvanceMed Research, Lawrenceville, New Jersey
  - Carolina Clinical Trials, LLC, Concord, North Carolina
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Seattle Urology Research Center, Burien, Washington
- Austria (2):
  - AKH Linz GmbH, Department of Urology, Linz, Upper Austria
  - Universitätsklinik für Urologie und Andrologie, Landeskrankenhaus Salzburg (University hospital for Urology and Andrology), Salzburg
- Czechia (3):
  - Thomayerova nemocnice Urologické oddělení, Prague, Praha 4 - Krč
  - University Hospital Hradec Králové, Hradec Králové
  - University Hospital Olomouc, Olomouc
- Universitätsklinikum RWTH Aachen, Klinik für Urologie, Aachen, North Rhine-Westphalia, Germany
- Lithuania (3):
  - PI Hospital of Lithuanian University of Health Sciences, Kauno Klinikos, Kaunas
  - PI Klaipėda University Hospital, Klaipėda
  - PI Vilnius University Hospital, Santariškių Klinikos, Vilnius
- Poland (4):
  - Centralny Szpital Kliniczny MSW w Warszawie, Klinika Urologii i Urologii Onkologicznej, Warzawa, Warzawa
  - Centrum Onkologii - Instytut im. Marii Skłodowskiej-Curie Klinika Nowotworów Układu Moczowego, Warzawa, Warzawa
  - Uniwersyteckie Centrum Kliniczne, Klinika Urologii, Gdansk
  - "DERMED" Centrum Medyczne Sp. z o.o., Lodz
- Slovakia (2):
  - UROCENTRUM MILAB, s.r.o., Prešov
  - Fakultná nemocnica s poliklinikou Žilina Urológia, Žilina
- Taiwan (6):
  - Kaohsiung Veteran General Hospital (VGHKS), Kaohsiung City, Pingtung
  - China Medical University Hospital (CMUH), Taichung, Taichung
  - Taichung Veteran General Hospital (VGHTC), Taichung, Taichung
  - National Cheng Kung University Hospital (NCKUH), Tainan, Tainan
  - National Taiwan University Hospital (NTUH), Taipei City, Taipei
  - Chang Gung Memorial Hospital, LinKou (CGMH-LK), Taoyuan

RESULTS

PARTICIPANT FLOW:
Groups:
- Leuprolide Mesylate 50mg: All subjects were males with advanced prostate carcinoma. They were injected twice with a depot formulation containing 50 mg of Leuprolide Mesylate. The first dose on day 0 the second dose on day 168 (six months apart). Subjects were followed until day 336.
  Leuprolide Mesylate: Subcutaneous injection of 50mg Leuprolide Mesylate
Period: Overall Study
Arm/Group | Leuprolide Mesylate 50mg
Started | 137
ITT | 137
PP | 124
PK Subgroup | 31
Completed | 122
Not Completed | 15

BASELINE CHARACTERISTICS:
Arm/Group | Leuprolide Mesylate 50mg
Number analyzed (Participants) | 137
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.1 (8.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 137
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 61
  Unknown or Not Reported | 73
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 123
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Austria | 1
  United States | 64
  Czechia | 17
  Taiwan | 2
  Poland | 5
  Slovakia | 18
  Lithuania | 29
  Germany | 1

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Leuprolide Mesylate (LMIS 50mg)
Description: The percentage of subjects with a serum testosterone concentration suppressed to castrate levels (≤ 50 ng/dL) following the first injection of LMIS 50 mg from Day 28 through Day 336 (remaining duration of the study).
Time Frame: baseline to 28 days, 28 days to 336 days
Population: ITT
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Leuprolide Mesylate 50mg
Number analyzed (Participants) | 137
percentage of participants | 97.0 [92.2 to 98.9]

2. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: Safety analysis was based on the safety information from the laboratory evaluations, AEs, and SAEs.
Time Frame: 336 days
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Leuprolide Mesylate 50mg
Number analyzed (Participants) | 137
Participants
  TEAE | 114
  Drug-related AEs | 85
  SAE | 20

ADVERSE EVENTS:
Time Frame: 336 days
Arm/Group | Leuprolide Mesylate 50mg
All-Cause Mortality (participants affected / at risk) | 3/137
Serious Adverse Events (participants affected / at risk) | 20/137
Other Adverse Events (participants affected / at risk) | 114/137
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Leuprolide Mesylate 50mg (N=137)
Angina pectoris (Cardiac disorders) | 1 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Death (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Bronchitis bacterial (Infections and infestations) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1)
Intermittent claudication (Vascular disorders) | 1 (1)
Peripheral artery occlusion (Vascular disorders) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Leuprolide Mesylate 50mg (N=137)
Fatigue (General disorders) | 9 (10)
Injection site pain (General disorders) | 10 (13)
Nasopharyngitis (Infections and infestations) | 7 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (12)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 (18)
Nocturia (Renal and urinary disorders) | 8 (9)
Hot flush (Vascular disorders) | 67 (69)
Hypertension (Vascular disorders) | 20 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All information from the trial is property of the Sponsor and the PI has no right on it except the prior writing authorization of the sponsor.